CLINICAL TRIAL: NCT00874185
Title: Satisfaction With Treatment In Patients With Erectile Dysfunction And Cardiovascular Risk And/Or Previous Cardiovascular Event.
Brief Title: Satisfaction With Phosphodiesterase 5 Inhibitors Treatment In Patients With Cardiovascular Risk
Acronym: TIERRA
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481256; A1481256
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
Keywords: satisfaction
MeSH Terms: conditions — Erectile Dysfunction; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire: filling in questionnaires

SUMMARY:
Evaluate satisfaction in people treated with IPDE5 inhibitors over time

DETAILED DESCRIPTION:
12 first patients that are eligible

ELIGIBILITY:
Inclusion Criteria:

* CV risk factors
* Male above 18

Exclusion Criteria:

* Non-informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with cv risk
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2007-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
EDITS | 6 months
SEAR | 6 months

SECONDARY OUTCOMES:
Medication prescribed | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481256&StudyName=Satisfaction%20With%20IPDE5%20Treatment%20In%20Patients%20With%20CV%20Risk